CLINICAL TRIAL: NCT00695565
Title: A Multicenter, Randomized, Double-Blind, Parallel-Group Study Comparing the Efficacy and Safety of Clonidine Topical Gel, 0.1% With Placebo in the Management of Pain Associated With Painful Diabetic Neuropathy
Brief Title: Efficacy and Safety Study of ARC-4558 for Management of Pain Associated With Painful Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arcion Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLO-027
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Results first posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-09

CONDITIONS: Painful Diabetic Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo Gel (Placebo Comparator): Placebo Gel is vehicle without clonidine
  Interventions: Drug: Placebo Gel
- Clonidine Topical Gel (ARC-4558) (Active Comparator): Clonidine Topical Gel contains 0.1% clonidine hydrochloride
  Interventions: Drug: Clonidine Topical Gel (ARC-4558)

INTERVENTIONS:
Drug: Placebo Gel — TID x 12 weeks
  Arms: Placebo Gel
Drug: Clonidine Topical Gel (ARC-4558) — TID x 12 weeks
  Arms: Clonidine Topical Gel (ARC-4558)

SUMMARY:
The purpose of this study is to determine whether ARC-4558 is effective in managing pain associated with painful diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* has Type 1 or Type 2 diabetes mellitus
* has a history of chronic pain attributable to a symmetrical stocking distribution neuropathy in the lower extremities for a duration of at least six months but less than or equal to five years prior to Screening

Exclusion Criteria:

* has neuropathy secondary to non-diabetic causes
* has a significant neurological disorder or a condition that can cause symptoms that mimic peripheral neuropathy or might confound assessment of PDN
* has other chronic pain with intensity at or greater than the bilateral pain in the feet/toes
* is using an implanted medical device (eg, spinal cord stimulator, intrathecal pump, or peripheral nerve stimulator) for the treatment of pain
* is pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2008-05; Primary Completion 2009-12 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James N Campbell, M.D., Study Chair — Arcion Therapeutics Inc
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, School of Medicine, Birmingham, Alabama
  - Northern California Research, Sacramento, California
  - Neurological Research Institute, Santa Monica, California
  - Metabolic Research Institute, West Palm Beach, Florida
  - Pain Treatment Center of the Bluegrass, Lexington, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Massachuetts Medical School, Division of Diabetes- Clinical Research Office, Worcester, Massachusetts
  - The Creighton Diabetes Center, Omaha, Nebraska
  - University of Rochester Medical Center, Rochester, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Waccamaw Pain Partners/Crescent Moon Research, Murrells Inlet, South Carolina
  - The Nerve and Muscle Center of Texas, Houston, Texas
  - Diabetes and Glandular Disease Center, San Antonio, Texas
  - Strelitz Diabetes Institute, Eastern Virginia Medical School, Norfolk, Virginia
  - Swedish Pain Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Campbell CM, Kipnes MS, Stouch BC, Brady KL, Kelly M, Schmidt WK, Petersen KL, Rowbotham MC, Campbell JN. Randomized control trial of topical clonidine for treatment of painful diabetic neuropathy. Pain. 2012 Sep;153(9):1815-1823. doi: 10.1016/j.pain.2012.04.014. Epub 2012 Jun 8. PMID 22683276
- [Derived] Serednicki WT, Wrzosek A, Woron J, Garlicki J, Dobrogowski J, Jakowicka-Wordliczek J, Wordliczek J, Zajaczkowska R. Topical clonidine for neuropathic pain in adults. Cochrane Database Syst Rev. 2022 May 19;5(5):CD010967. doi: 10.1002/14651858.CD010967.pub3. PMID 35587172

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from May 2008 until September 2009. All study sites were medical clinics.
Pre-assignment Details: Subjects were required to meet all eligibility criteria at both the Screening and Baseline visits. If a subject met the Screening criteria but not the Baseline criteria, the subject was not eligible for enrollment.
  Two subjects were randomized but were not treated because they were found ineligible. They are not counted in the 180 enrolled.
Period: Overall Study
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Started | 90 | 90
Completed | 77 | 81
Not Completed | 13 | 9
Not completed — Lost to Follow-up | 4 | 4
Not completed — Adverse Event | 3 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 1 | 1
Not completed — Subject did not follow instructions | 1 | 1

BASELINE CHARACTERISTICS:
Population: ITT (Intent-to-Treat)
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558) | Total
Number analyzed (Participants) | 90 | 90 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (9.5) | 59.4 (9.9) | 58.5 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 46 | 94
  Male | 42 | 44 | 86
Region of Enrollment [Number; unit: participants]
  United States | 90 | 90 | 180

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Average Daily Pain NPRS (Numeric Pain Rating Scale) Score; mLOCF Imputation
Description: Pain in the feet was scored daily at bedtime by the subject on a 0-10 numeric pain rating scale (NPRS) through Day 84. Subjects were asked to record average pain in the feet over the past 24 hours. A score of 0 indicated "no pain" and a score of 10 was "worst possible pain".
  The change in pain is represented as Week 12 minus Baseline, so greater negative numbers represent more improvement (more pain relief).
Time Frame: Baseline (average of Days -7 to -1) and Week 12 (Average of Days 78 to 84)
Population: One treated subject had no recorded scores and could not be included. Imputation was mLOCF (modified Last Observation Carried Forward): LOCF for subjects who discontinued early, except if withdrawal was associated with an adverse event (AE) potentially related to study medication (in which case Baseline Observation Carried Forward (BOCF) was used).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Gel: Placebo Gel is vehicle without clonidine; Subjects applied the gel to their feet 3 times daily starting on Day 1.
- Clonidine Topical Gel (ARC-4558): Clonidine Topical Gel contains 0.1% clonidine hydrochloride; Subjects applied the gel to their feet 3 times daily starting on Day 1.
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale
  All subjects | -1.9 (1.9) | -2.4 (2.1)
  Capsaicin response ≥ 2 | -1.5 (1.8) | -2.7 (1.9)
Statistical Analysis 1: Comparison: Placebo Gel vs Clonidine Topical Gel (ARC-4558); This analysis does not take into account the subjects' screening capsaicin response (measure of nociceptor function); Test type: Superiority or Other; p = 0.168, Mixed Models Analysis; Mean Difference (Net) = -0.5
Statistical Analysis 2: Comparison: Placebo Gel vs Clonidine Topical Gel (ARC-4558); Each subject was screened for responsiveness of nociceptors in the skin to a capsaicin stimulus (rated on 0-10 pain scale; 0=no pain and 10=worst possible pain). The interaction term composed of treatment assignment and capsaicin threshold was examined at the prespecified alpha level of 0.1. This analysis includes subjects with a capsaicin rating of ≥ 2. Thirty (30) subjects in the Placebo group and 33 subjects in the active Clonidine Topical Gel (ARC-4558) group had capsaicin scores ≥ 2; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis; Mean Difference (Net) = -1.2

2. Secondary Outcome: Change From Baseline in Average Daily Pain NPRS Score for Each Week of Treatment; mLOCF Imputation
Description: Pain in the feet was scored daily at bedtime by the subject on a 0-10 numeric pain rating scale (NPRS). Subjects were asked to record average pain in the feet over the past 24 hours. A score of 0 indicated "no pain" and a score of 10 was "worst possible pain". A weekly average was calculated from the daily scores for each week. The change in pain is represented as the average weekly score minus Baseline, so greater negative numbers represent more improvement (more pain relief).
Time Frame: Baseline (average of Days -7 to -1) and Weeks 1 through 12 (weekly averages)
Population: One treated subject had no recorded scores and could not be included. Imputation was a modified LOCF (LOCF for subjects who discontinued early, except if withdrawal was associated with an adverse event (AE) potentially related to study medication, in which case BOCF was used). Additional BOCF analyses have been published (Pain 2012, see citation)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale
  Week 1 | -0.6 (1.01) | -0.7 (1.34)
  Week 2 | -1.0 (1.30) | -1.0 (1.45)
  Week 3 | -1.2 (1.47) | -1.5 (1.58)
  Week 4 | -1.5 (1.63) | -1.6 (1.71)
  Week 5 | -1.7 (1.77) | -1.7 (1.65)
  Week 6 | -1.8 (1.84) | -1.8 (1.74)
  Week 7 | -1.8 (1.83) | -2.1 (1.86)
  Week 8 | -1.9 (1.93) | -2.2 (1.92)
  Week 9 | -1.9 (1.96) | -2.3 (1.95)
  Week 10 | -1.9 (1.98) | -2.4 (2.06)
  Week 11 | -1.9 (1.93) | -2.3 (2.12)
  Week 12 | -1.9 (1.91) | -2.4 (2.12)

3. Secondary Outcome: Change From Baseline to Week 12 in the Worst Daily Pain NPRS Score; mLOCF Imputation
Description: Pain in the feet was scored daily at bedtime by the subject on a 0-10 numeric pain rating scale. Subjects were asked to record the worst pain in their feet over the past 24 hours. A score of 0 indicated "no pain" and a score of 10 was "worst possible pain". The change in pain is represented as Week 12 minus Baseline, so greater negative numbers represent greater improvement (greater pain relief).
Time Frame: Baseline (average of Days -7 to -1) and Week 12 (average of Days 78 to 84)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -2.1 (2.1) | -2.5 (2.3)

4. Secondary Outcome: Percentage of Subjects Who Experience at Least 30% Reduction in Average Daily Pain From Baseline; mLOCF Imputation
Description: Pain in the feet was scored daily at bedtime by the subject on a 0-10 numeric pain rating scale (NPRS). Subjects were asked to record average pain in the feet over the past 24 hours. A score of 0 indicated "no pain" and a score of 10 was "worst possible pain".
Time Frame: Baseline (average of Days -7 to -1) and Week 12 (average of Days 78 to 84)
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
percentage of subjects | 47 | 52

5. Secondary Outcome: Percentage of Subjects Who Experience at Least 50% Reduction in Average Daily Pain From Baseline; mLOCF Imputation
Description: as for outcome 4
Time Frame: Baseline (average of Days -7 to -1) and Week 12 (average of Days 78 to 84)
Population: as for outcome 2
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
percentage of subjects | 32 | 37

6. Secondary Outcome: Change From Baseline in the Brief Pain Inventory (BPI) Severity Scale at Week 12; mLOCF Imputation
Description: The Brief Pain Inventory was completed by the subject at clinic visits. The Severity Scale (of 0 to 40) is a composite score, which is the sum of the individual ratings for worst pain, least pain, average pain, and current pain. Each individual question is rated on a scale of 0 to 10, where 0 indicates "No Pain" and 10 indicates "Pain as bad as you can imagine". The change in pain severity is represented as Week 12 minus Baseline, so greater negative numbers represent greater improvement (pain relief).
Time Frame: Baseline and Week 12
Population: One subject in the active Clonidine Gel group was lost to follow-up before Baseline pain scores were confirmed and before any post-baseline efficacy evaluations were performed. This subject was excluded from the efficacy analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -7.9 (8.5) | -9.6 (8.7)

7. Secondary Outcome: Change From Baseline in the Brief Pain Inventory Functional Interference Scale at Week 12; mLOCF Imputation
Description: The Brief Pain Inventory was completed by the subject at clinic visits. The Functional Interference Scale (of 0 to 70) is a composite score that measures the degree to which pain interferes with mood, walking, work, relationships, sleep, general activity, and enjoyment of life. The composite score is a sum of the seven individual question scores. Each individual question is rated in reference to pain over the past 24 hours on a scale of 0 to 10, where 0 indicates that pain "does not interfere" and 10 indicates that pain "completely interferes" with that function, so lower scores represent better outcomes on this scale.
  The change in functional interference is represented as Week 12 minus Baseline, so greater negative numbers represent more improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -15.1 (14.9) | -17.3 (17.5)

8. Secondary Outcome: Change From Baseline to Week 12 in Overall Quality of Sleep (Chronic Pain Sleep Inventory)
Description: Subjects rated overall quality of sleep over the past week using a 100 mm Visual Analog Scale (VAS) where 100=Excellent and 0=Very Poor. This scale was completed during clinic visits. Change from Baseline is a positive value where quality of sleep improved.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | 17.7 (33.4) | 19.2 (31.3)

9. Secondary Outcome: Change From Baseline to Week 12 in the Depression Score of the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS was completed at the Baseline and Week 12 clinic visits. The Depression Score component of the HADS includes 7 questions, each with 4 possible answer choices (rated 0 to 3). The composite score is created by adding the scores of the 7 individual questions. A score of 0 to 7 is Normal, 8-10 indicates Mild Depression, 11-14 indicates Moderate Depression, and 15-21 indicates Severe Depression. The change from Baseline is calculated as the Week 12 composite score minus the Baseline composite score.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -0.4 (2.6) | -0.9 (2.3)

10. Secondary Outcome: Change From Baseline to Week 12 in the Anxiety Score of the Hospital Anxiety and Depression Scale (HADS)
Description: The HADS was completed at the Baseline and Week 12 clinic visits. The Anxiety Score component of the HADS includes 7 questions, each with 4 possible answer choices (rated 0 to 3). The composite score is created by adding the scores of the 7 individual questions. A score of 0 to 7 is Normal, 8-10 indicates Mild Anxiety, 11-14 indicates Moderate Anxiety, and 15-21 indicates Severe Anxiety. The change from Baseline is calculated as the Week 12 composite score minus the Baseline composite score.
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -0.6 (2.67) | -1.1 (3.14)

11. Secondary Outcome: Change From Baseline to Week 12 in the McGill Pain Questionnaire (Short Form) Total Score
Description: The McGill Pain Questionnaire asks subjects to rate 15 different kinds of pain, each on a scale of 0 to 3 (0=None, 1=Mild, 2=Moderate, 3=Severe). The total score is a sum of the individual ratings and has a range from 0 to 45, where higher numbers indicate more pain. The 15 types of pain assessed are throbbing, shooting, stabbing, sharp, cramping, gnawing, hot-burning, aching, heavy, tender, splitting, tiring-exhausting, sickening, fearful, and punishing-cruel. This scale was completed at the Baseline and Week 12 clinic visits. The change from Baseline is calculated as the Week 12 total score minus the Baseline total score, so greater negative numbers indicate more improvement (pain relief).
Time Frame: Baseline and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 89
units on a scale | -7.3 (8.3) | -8.7 (9.8)

12. Secondary Outcome: Patient Global Impression of Change (PGIC) at Week 12
Description: At Week 12 the subject was asked to rate their total improvement relative to Baseline, whether or not, in their judgement, it was due entirely to study drug treatment or not. Answer choices were: (+3) very much improved, (+2) much improved, (+1) minimally improved, (0) no change, (-1) minimally worse, (-2) much worse, (-3) very much worse.
Time Frame: Week 12
Population: All subjects with a PGIC score were analyzed.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 85 | 85
percentage of subjects
  Very Much Improved | 11.8 | 21.2
  Much Improved | 32.9 | 27.1
  Minimally Improved | 31.8 | 28.2
  No Change | 21.2 | 22.4
  Minimally Worse | 1.2 | 1.2
  Very Much Worse | 1.2 | 0

13. Secondary Outcome: Clinician Global Impression of Change (CGIC) at Week 12
Description: At Week 12, the Investigator was asked to independently rate the subject's total improvement relative to Baseline, whether or not, in their judgement, it was due entirely to study drug treatment or not. Answer choices were: (+3) very much improved, (+2) much improved, (+1) minimally improved, (0) no change, (-1) minimally worse, (-2) much worse, (-3) very much worse.
Time Frame: Week 12
Population: All subjects with a CGIC score were analyzed.
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 85 | 86
percentage of subjects
  Very Much Improved | 5.8 | 16.5
  Much Improved | 38.4 | 30.6
  Minimally Improved | 27.9 | 24.7
  No Change | 25.6 | 27.1
  Minimally Worse | 2.3 | 1.2
  Very Much Worse | 0 | 0

14. Secondary Outcome: Change in Blood Pressure From Baseline to Week 12
Description: Systolic and Diastolic Blood Pressure were measured at clinic visits. This outcome assesses the change in blood pressure from Baseline to Week 12 of treatment.
Time Frame: Baseline and Week 12
Population: ITT (Intent-to-Treat)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Number analyzed (Participants) | 90 | 90
mmHg
  Change in Systolic BP | -0.4 (20.6) | 1.0 (13.9)
  Change in Diastolic BP | -0.2 (9.4) | 1.0 (8.8)

ADVERSE EVENTS:
Arm/Group | Placebo Gel | Clonidine Topical Gel (ARC-4558)
Serious Adverse Events (participants affected / at risk) | 3/90 | 3/90
Other Adverse Events (participants affected / at risk) | 28/90 | 19/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Gel (N=90) | Clonidine Topical Gel (ARC-4558) (N=90)
Acute Coronary Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Abscess Neck (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Gel (N=90) | Clonidine Topical Gel (ARC-4558) (N=90)
Headache (Nervous system disorders) | 10 | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 7 | 3
Pain (General disorders) | 6 | 0
Nasopharyngitis (Infections and infestations) | 4 | 5
Toothache (Gastrointestinal disorders) | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may not publish or present any study information without the express written approval of the Sponsor. The Sponsor may withhold approval for publication or presentation.